CLINICAL TRIAL: NCT02833324
Title: Can a Fitbit (a Mobile Tracking Device) Increase Ambulation of Colorectal Surgical Patients in the Postoperative Period?
Brief Title: Fitbit for Postoperative Ambulation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Emory University (Other)
Responsible Party: Principal Investigator, Patrick Sean Sullivan MD, MD, Emory University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: IRB00088864
Record Dates: First submitted 2016-07-12; First posted 2016-07-14 (Estimated); Last update posted 2017-10-17 (Actual); Status verified 2017-10

CONDITIONS: Postoperative Care
Keywords: Postoperative Period; Colorectal Surgery; Surgery

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Fitbit with ambulation reminder alarms (Experimental): Study participants who are postoperative for colorectal surgery will wear a Fitbit (a wireless activity tracking device) to count steps taken during their postoperative hospitalization. In addition to being educated on the importance of postoperative ambulation, this arm will have 5 alarms every day reminding them to ambulate.
  Interventions: Behavioral: Education regarding ambulation; Behavioral: Ambulation reminder alarms; Other: Fitbit
- Fitbit without ambulation reminder alarms (Active Comparator): Study participants who are postoperative for colorectal surgery will wear a Fitbit (a wireless activity tracking device) to count steps taken during their postoperative hospitalization. Participants will be educated on the importance of postoperative ambulation but will not have ambulation reminder alarms.
  Interventions: Behavioral: Education regarding ambulation; Other: Fitbit

INTERVENTIONS:
Behavioral: Education regarding ambulation — The participants will be educated on the importance of postoperative ambulation during the recovery period.
Behavioral: Ambulation reminder alarms — Participants in the intervention arm will receive 5 daily alarms to prompt them to ambulate. Alarms will be set to ring at 9am, 11am, 2pm, 5pm and 9pm. The Fitbit will be worn from the day of surgery (postoperative day 0) through postoperative day 9 or hospital discharge, whichever occurs first.
  Arms: Fitbit with ambulation reminder alarms
Other: Fitbit — Participants who are postoperative for colorectal surgery, who have been cleared to ambulate during recover, will be equipped with an off-the-shelf Fitbit device (a wireless activity tracking device) which will record steps taken while the participant is hospitalized. The Fitbit will be worn from the day of surgery (postoperative day 0) through postoperative day 9 or hospital discharge, whichever occurs first.

SUMMARY:
This trial will investigate whether using reminder alarms with a wireless activity tracking device (Fitbit) will increase daily ambulation in individuals who have just had colorectal surgery.

DETAILED DESCRIPTION:
Early mobilization after surgery has been shown to reduce recovery time, incidence of venous thromboembolism, length of hospital stay and both pulmonary and general post-operative complications. Ambulation is also a main tenant of a fast-track recovery protocol known as Enhanced Recovery After Surgery (ERAS), which is commonly used among colorectal surgical practices and being implanted across other surgical practices. Despite evidence supporting its benefit, early ambulation has been identified as the one of the most difficult clinical interventions to enforce and to measure.

The primary objective of this trial is to investigate whether the use of wireless activity tracking device (Fitbit) with 5 daily reminder alarms will increase daily ambulation on postoperative day 0 until post operative day 9 or hospital discharge (whichever occurs first). Secondary objectives include evaluating the effect of Fitbit as a motivating factor on the frequency of postoperative ileus, time to return of bowel function, number of venous thromboembolism (VTE), pneumonia (PNA) and other pulmonary complications, number of code Medical Emergency Team (MET) alerts, and overall cost saving.

ELIGIBILITY:
Inclusion Criteria:

* Undergoing an elective surgical procedure in colorectal services at Emory University Hospital

Exclusion Criteria:

* Post-surgical admission into the intensive care unit (ICU)
* Have an open abdomen due to surgical complications
* Wound Vacuum Assisted Closure (VAC) dependent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 48 (Actual)
Dates: Start 2016-07; Primary Completion 2016-12 (Actual); Study Completion 2016-12 (Actual)

PRIMARY OUTCOMES:
Comparison of number of steps taken between study arms | Up to 10 days (postoperative day 0 through postoperative day 9)
  The number of steps taken by each participant will be measured by a Fitbit, which is a wireless activity tracking device. The number of steps taken will be compared between the study arm receiving the ambulation reminder alarms and the study arm without reminder alarms. The Fitbit is commercially available and is worn on the wrist. Data will be collected from the Fitbit wirelessly using a dedicated study data collection phone and linked with an anonymized patient identifier. Data collection phones attached to chargers will be placed in patient rooms within range of the hospital bed to enable automatic wireless data collection.

SECONDARY OUTCOMES:
Comparison of time to first ambulation between study arms | Up to 10 days (postoperative day 0 through postoperative day 9)
  The duration of time from administration of the Fitbit device until first postoperative ambulation will be compared between the study arm receiving the ambulation reminder alarms and the study arm without reminder alarms. Participants cleared to ambulate will be given a package containing the Fitbit device, paired study phone, and chargers while in the Post Anesthesia Care Unit (PACU). Participants will be instructed to equip the device prior to discharge from the PACU.
Comparison of incidence of prolonged postoperative ileus between study arms | Up to 10 days (postoperative day 0 through postoperative day 9)
  The incidence of prolonged postoperative ileus during hospitalization will be compared between the study arm receiving the ambulation reminder alarms and the study arm without reminder alarms.
  For this study, postoperative ileus is defined as the interval from surgery until there is passage of flatus or stool and an oral diet is tolerated. Prolonged postoperative ileus is determined to be present if two or more of the following criteria are met on or after postoperative day 4, without prior resolution of postoperative ileus:
  * Nausea or vomiting
  * The inability to tolerate an oral diet over 24 hours
  * Absence of flatus over 24 hours
  * Abdominal distension
  * Radiologic confirmation
Comparison of incidence of pulmonary complications between study arms | Up to 10 days (postoperative day 0 through postoperative day 9)
  The incidence of pulmonary complications during hospitalization will be compared between the study arm receiving the ambulation reminder alarms and the study arm without reminder alarms. For this study, pulmonary complications are defined as respiratory failure requiring mechanical ventilation, pneumonia, atelectasis requiring bronchoscopic intervention, or pneumothorax or pleural effusion requiring percutaneous intervention.
Comparison of incidence of venous thromboembolism between study arms | Up to 10 days (postoperative day 0 through postoperative day 9)
  The incidence of venous thromboembolism occurring during hospitalization will be compared between the study arm receiving the ambulation reminder alarms and the study arm without reminder alarms. Venous thromboembolism is when a blood clot (thrombus) forms within a vein and includes deep vein thrombosis (DVT) and pulmonary embolism (PE).
Comparison of length of postoperative hospital stay between study arms | Up to 10 days (postoperative day 0 through postoperative day 9)
  The length of hospitalization following surgery will be compared between the study arm receiving the ambulation reminder alarms and the study arm without reminder alarms.

CONTACTS AND LOCATIONS:
Overall Officials: Patrick S Sullivan, MD, Principal Investigator — Emory University
Locations (1):
- Emory University Hospital, Atlanta, Georgia, United States

IPD SHARING:
Plan to Share IPD: No